CLINICAL TRIAL: NCT01868711
Title: Psychological Mindedness as a Predictor of Success in Cognitive Behavior Therapy for Depressed Patients
Brief Title: Cognitive Behavior Therapy for Depression
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ronit Kishon, Associate Professor of Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6806R; R21MH121915-01A1 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-06-04 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Depression
Keywords: Cognitive Behavior Therapy; Self-awarness; Supportive Therapy; Virtual psychotherapy
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Depressed patients will be randomized between cognitive behavor therapy and supportive therapy.
Oversight: Data Monitoring Committee: No

ARMS (2):
- *Cognitive behavior therapy (Active Comparator): Depressed patients will receive 12 virtual sessions of cognitive behavior therapy (CBT) for depression. CBT Includes behavior activation, correcting distorted thoughts, and other tools to reduce symptoms.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Supportive psychotherapy (Other): Supportive psychotherapy aims to strengthen the patient's ability to cope effectively with various life stressors. Specifically, in our study, supportive psychotherapy will be geared towards reducing or alleviating symptoms of depression. The sessions will be administered virtually.
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy
  Other Names: Supportive psychotherapy

SUMMARY:
Psychological mindedness(PM) is a metacognitive process in which the person uses his cognitive and affective abilities to understand his thoughts, feelings, and his behaviors as they interact with his internal experiences and his external experiences in the world. It dynamically modifies his behavior to move towards self-actualization in a manner positive to himself and the world. We investigate whether the assessment of PM can distinguish depressed patients who benefit from CBT.

DETAILED DESCRIPTION:
Cognitive Behavior Therapy (CBT) is one of the most effective psychotherapy for depression. Yet, it is effective only for 40% of the depressed people who receive this treatment. Currently, there is no method of predicting who can be helped among depressed patients by CBT. In this study, we examine whether the level of psychological mindedness can predict who may benefit from CBT among depressed patients.

Participants who are clinically depressed are randomized to 12 sessions of CBT and supportive therapy. The evaluation process and all sessions will be administered virtually using HIPAA-compliant video teleconferencing. Participants must have access to the internet and have video conferencing capabilities. Besides the virtual sessions, participants will need to come in person once for a urine & blood test (protocol #6669) and twice for an electroencephalogram (EEG) (protocol #6559). Dr. Jürgen Kayser who is heading the EEG lab is a co-PI on this grant.

Please exercise caution when traveling in public and follow public health guidelines, such as wearing masks in public and avoiding crowds. It would be best if you stay informed of public health recommendations and guidelines regarding COVID-19, such as those issued by the Centers for Disease Control (CDC.gov) and local governments. If you have questions about how you will travel for appointments or do not feel safe traveling, please let us know, and know that you can call to reschedule visits.

It is important to note that subjects who enroll in the study can't take any psychiatric medications, nor can they attend any other psychotherapy besides what is offered in the study. Should the participant decide to make alternations and use medication, this will not affect their participation in psychotherapy or this study.

Participants who are eligible for the study will begin within two weeks after the evaluation visit. An evaluator will rate the HDRS-17 and CG I-Severity. If they are still eligible, they will sign the study consent form, have the study explained, including its risks and possible benefits, as well as alternatives and its voluntary nature. Once they sign the consent form, patients will complete a battery of self-report instruments online. Also, they will be interviewed by a clinician with a structured clinical interview of PM. They will then be randomized between CBT and supportive therapy (control group) and will schedule their weekly virtual sessions with the study therapist. During 12 weeks, they will be clinically monitored by Beck Depression Inventory at the beginning of every session and HDRS-17 every three weeks. They will complete study measures at week six and after the 12 weeks sessions.

Study participants who do not remit (end treatment HDRS-17 > 7) at the end of the CBT trial will receive a referral for alternative psychotherapy per the patient's preference.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 65 (inclusive).
* Primary DSM-IV-TR diagnosis of major depression
* A negative urine toxicology, i.e., a urine specimen that does not test positive for the use of drugs of abuse or use of benzodiazepines.
* Ability to give informed consent.
* Fluent in English

Exclusion Criteria:

* Patients who have a "lifetime" history of Schizophrenia or other current psychotic disorder, Major Depressive Disorder with Psychotic or Catatonic features, Bipolar I Affective Disorder, or Organic Mental Disease.
* DSM-V substance abuse or dependence within the past 6 months (except nicotine or caffeine).
* Active suicidal or homicidal ideation, or judged to be at serious suicide risk.
* Any unstable medical or neurological condition.
* Presently receiving psychotherapy or psychotropic medications.
* Prior History of CBT for Depression treatment failure.
* Left-handedness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Level of depression as measured by the Hamilton Depression Rating Scale | Up to 12 weeks.
  Outcome measure of depression will be assessed as the change in depression between baseline (pre-treatment) and post treatment (up to 12 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Kishon, Ph.D., Principal Investigator — New York State Psychiatric Institute, Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about the study — http://depression-nyc.org

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT01868711/Prot_SAP_ICF_001.pdf